CLINICAL TRIAL: NCT05481190
Title: The Impact Of A Tele-Exercise Program For Children With Cystic Fibrosis During The Covid-19 Pandemic On Quality Of Life: A Randomized Controlled Trial
Brief Title: The Impact Of A Tele-Exercise Program For Children With Cystic Fibrosis During The Covid-19 Pandemic On Quality Of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Merve Koyun, Principal Investigator, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Tele-Exercise
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Cystic Fibrosis; Exercise Addiction; Nursing Caries; Quality of Life; Exercise Adherence
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: The study is a randomized controlled experimental study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-exercise program to Child with Cystic Fibrosis (Experimental): Inclusion criteria were "Voluntary to participate in the study", "Getting consent from parents", "Being a child with cystic fibrosis between the ages of 10-18", "Having no psychological health problems", "No physical problems that would prevent the child from exercising" and "Computer/ owning a smart phone and being able to use these devices", "Having an internet connection at home".
  The exclusion criteria were "Not volunteering to participate in the study", "Not being able to get consent from their parents", "Being under the age of 10 or over the age of 18 with a diagnosis of Cystic Fibrosis", "Having a psychological health problem", "Having a physical problem that prevents the child from exercising" and "Not having a computer/smart phone and not being able to use these devices" and "Not having an internet connection at home".
  Exclusion criteria are "Not participating in the exercise regularly (at least 2 times)", "Not wanting to continue working out".
  Interventions: Behavioral: Tele-Exercise Program; Behavioral: Just observation
- Without exercise Child with Cystic Fibrosis (Experimental): Inclusion criteria were "Voluntary to participate in the study", "Getting consent from parents", "Being a child with cystic fibrosis between the ages of 10-18", "Having no psychological health problems", "No physical problems that would prevent the child from exercising" and "Computer/ owning a smart phone and being able to use these devices", "Having an internet connection at home".
  The exclusion criteria were "Not volunteering to participate in the study", "Not being able to get consent from their parents", "Being under the age of 10 or over the age of 18 with a diagnosis of Cystic Fibrosis", "Having a psychological health problem", "Having a physical problem that prevents the child from exercising" and "Not having a computer/smart phone and not being able to use these devices" and "Not having an internet connection at home".
  Exclusion criteria are "Not participating in the exercise regularly (at least 2 times)", "Not wanting to continue working out".
  Interventions: Behavioral: Tele-Exercise Program; Behavioral: Just observation

INTERVENTIONS:
Behavioral: Tele-Exercise Program — Data collection tools were applied to the tele-exercise group and control group at the beginning of the study. For the tele-exercise group, by the researcher, Exp. A 6-week exercise program was created under the consultancy of a physiotherapist. Children who met the research criteria were asked to do these exercises for 20 minutes, 3 times a week for 6 weeks. The exercises were performed online with the researcher at the scheduled time one day a week, and by the children twice a week. On the days they exercised, diaries consisting of semi-structured questions were sent to the children's addresses by cargo and they were allowed to keep a diary. Phone calls were made once a week to provide motivation and increase compliance with exercise. A smart watch was sent to the children by cargo to increase motivation. The children were asked to fill in the follow-up form, which was sent via weekly google forms.
Behavioral: Just observation — Standard care was given to the children in the control group.

SUMMARY:
The aim of this study was to examine the effect of the tele-exercise program applied to children with cystic fibrosis in the Covid-19 pandemic on the quality of life and the symptoms experienced during exercise

DETAILED DESCRIPTION:
Cystic fibrosis is a chronic, progressive, life-shortening, genetic, complex disease that affects multiple organs and systems. The care and treatment process of cystic fibrosis disease requires a multidisciplinary approach. Regular exercise (as it is an important component of therapeutic treatment) improves respiratory function in children with cystic fibrosis. However, the treatment burden of the disease in the child and the serious respiratory system complications caused by the Covid-19 infection during the pandemic process cause patients with cystic fibrosis to be in the high risk group. Since it is thought that it is difficult for children with cystic fibrosis to exercise during the pandemic process, home exercise programs have gained importance. With the developing technology, patients are consulted remotely, training and consultancy services are provided and they can be followed continuously through phone calls and video conferences. Nurses are an important part of the multidisciplinary team responsible for the protection, development and maintenance of the health of the individual in every period of life. They have assumed the roles of educator, consultant, decision-maker, therapeutic, caregiver and researcher in order to protect the quality of life of children with exercise programs and to ensure that they lead an active life. In order for nurses to make exercise a part of the lives of children with cystic fibrosis, they should determine the knowledge level, awareness and needs of children and their families, and provide adequate and effective counseling so that they can meet their individual needs.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary to participate in the study
* Getting consent from parents
* Being a child with cystic fibrosis between the ages of 10-18
* Having no psychological health problems
* No physical problems that would prevent the child from exercising"
* Computer/ owning a smart phone and being able to use these devices and having an internet connection at home".

Exclusion Criteria:

* Not participating in the exercise regularly (at least 2 times)",
* Not wanting to continue working out".
* Not being willing to participate in the study
* Not being able to get consent from their parents
* Being under the age of 10, over the age of 18 with a diagnosis of Cystic Fibrosis
* Having a psychological health problem
* Having a physical problem that prevents the child from exercising
* Using a computer/smartphone not having and not being able to use these devices
* Not having an internet connection at home".

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
changing the quality of life | Up to Six Weeks
  changing the quality of life of children with cystic fibrosis after tele-exercise program
affects the symptoms | Up to Six Weeks
  affects the symptoms experienced by the children in the tele-exercise group during exercise.

SECONDARY OUTCOMES:
changing the quality of life "Cystic Fibrosis Quality of Life Questionnaire" | Up to Six Weeks
  The questionnaire prepared in a four-point likert type is scored according to frequency and difficulty level or whether the answers are correct or incorrect. It is thought that the higher the total score obtained from the questionnaire, the higher the health-related quality of life.
affects the symptoms during the tele-exercise | Up to Six Weeks
  The children were asked to record their symptom findings daily and they were asked to share the recording documents with the researcher. In addition, the researcher questioned the symptom findings of the participants once a week by phone call and once a week via google form. The symptoms questioned through diary keeping, phone call and google form were recorded as symptom present/absent.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayıs University, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
other researhers may view the study once it is published.

REFERENCES:
- [Background] Chen JJ, Cooper DM, Haddad F, Sladkey A, Nussbaum E, Radom-Aizik S. Tele-Exercise as a Promising Tool to Promote Exercise in Children With Cystic Fibrosis. Front Public Health. 2018 Sep 28;6:269. doi: 10.3389/fpubh.2018.00269. eCollection 2018. PMID 30324099
- [Background] Cox NS, Alison JA, Button BM, Wilson JW, Holland AE. Feasibility and acceptability of an internet-based program to promote physical activity in adults with cystic fibrosis. Respir Care. 2015 Mar;60(3):422-9. doi: 10.4187/respcare.03165. Epub 2014 Nov 25. PMID 25425703
- [Result] Quittner AL, Buu A, Messer MA, Modi AC, Watrous M. Development and validation of The Cystic Fibrosis Questionnaire in the United States: a health-related quality-of-life measure for cystic fibrosis. Chest. 2005 Oct;128(4):2347-54. doi: 10.1378/chest.128.4.2347. PMID 16236893